CLINICAL TRIAL: NCT00970944
Title: A Multicenter Prospective Randomized Controlled Trial of the Effectiveness of Amantadine Hydrochloride in Promoting Recovery of Function Following Severe Traumatic Brain Injury
Brief Title: Effectiveness of Amantadine Hydrochloride for Treatment of Severe Traumatic Brain Injury (TBI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: JFK Medical Center (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joseph T Giacino, Director of Rehabilitation Neuropsychology, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H133A031713
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Rehabilitation; Disorders of Consciousness; Functional Outcome; Amantadine Hydrochloride
MeSH Terms: conditions — Brain Injuries, Traumatic; Consciousness Disorders | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amantadine HCL (Experimental): 100mg BID administered for 2 weeks, then increased to 150mg BID in week 3 if change on primary outcome measure (ie Disability Rating Scale, DRS) was less than 2 points after week 2. If change in DRS score remained less than 2 points after week 3, dose was increased to 200mg BID in week 4.
  Interventions: Drug: Amantadine Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine Hydrochloride — 184 patients who remain in VS or MCS 4 - 16 weeks post-TBI will be randomized in a stratified fashion to 4 weeks of amantadine (200 - 400 mg/day) followed by a 2-week washout period. The Disability Rating Scale (DRS) will be the primary dependent variable with the Coma Recovery Scale-Revised (CRS-R) serving as a supplementary measure.
  Other Names: Symmetrel
  Arms: Amantadine HCL
Drug: Placebo — Placebo administered twice daily.
  Arms: Placebo

SUMMARY:
This is a controlled trial of amantadine to improve level of function following severe traumatic brain injury.

The purpose of this study is:

1. To determine whether amantadine hydrochloride, given in a dose of 200-400 mg, improves functional recovery from the vegetative and minimally conscious states
2. To determine whether amantadine-related gains in function persist following drug discontinuation
3. To determine the safety profile of amantadine in patients with disorders of consciousness

DETAILED DESCRIPTION:
Severe traumatic brain injury may result in severe disorders of consciousness (DOC), including coma, the vegetative state (VS) and the minimally conscious state (MCS). The longer the duration of impaired consciousness, the worse the ultimate functional prognosis, with only about half of those individuals who remain unconscious for a month post-TBI regaining consciousness within a year. The severe functional disability associated with prolonged DOC places enormous emotional, financial, ethical, and logistical strains on caregivers and major resource demands on society. Numerous treatments have been recommended to hasten the return of consciousness or improve the ultimate level of recovery, including various psychotropic drugs, "coma stimulation" therapy and others. However, none of these treatments has proven efficacy in well-controlled research. The main obstacles to Class I evidence in this area have been the small samples of individuals with serious DOC in individual facilities, the variability of recovery trajectories within this heterogeneous population, and the reluctance to undertake placebo controlled trials.

In the proposed study, 7 facilities (including two with TBI Model Systems designations) that participated in a multi-center research network called the Consciousness Consortium, join with four additional brain injury rehabilitation centers (two in the U.S. and two in Europe) and a Data Coordinating Center at Columbia University, to conduct a prospective double blind randomized controlled trial of amantadine hydrochloride. 184 patients who remain in VS or MCS 4 - 16 weeks post-TBI will be randomized in a stratified fashion to 4 weeks of amantadine (200 - 400 mg/day) vs. placebo, followed by a 2-week washout period. The Disability Rating Scale (DRS) will be the primary dependent variable with the Coma Recovery Scale-Revised (CRS-R) serving as a supplementary measure. We hypothesize superior recovery in the amantadine group and maintenance of that advantage after washout. We will also explore whether treatment response differs by time post-injury and by diagnosis (i.e., VS or MCS) at treatment onset, and whether specific outcomes of importance to caregivers are achieved more often in the amantadine group. We have developed plans for intensive education of caregivers and clinicians about this study to address perceived barriers to enrollment and will also use the information gathered during these interactions to develop consumer-oriented dissemination activities. Project outputs and findings will be disseminated to appropriate consumer and professional audiences using a variety of formats and will include: (1) improved family member understanding of DOC which will facilitate improved adjustment and caregiving and (2) clear guidance to clinicians regarding the effectiveness of amantadine for persons with DOC.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between ages 16 and 65 with traumatic brain injury as defined by the TBI Model System syllabus (i.e., damage to brain tissue caused by an external mechanical force as evidenced by loss of consciousness or post-traumatic amnesia due to brain trauma, skull fracture, or objective neurological findings that can be reasonably attributed to TBI on physical or mental status examination).
* Individuals are at least 4 weeks but less than 16 weeks post-injury and have a Disability Rating Scale (DRS) score at enrollment of 12 or greater, and no consistent command following or functional communication (as defined by the JFK.

Exclusion Criteria:

* Women who are pregnant,
* Individuals with missile-type penetrating brain injury,
* Premorbid major CNS/developmental abnormality (e.g., mental retardation, prior significant brain damage, etc.),
* History of more than 1 seizure (clinical or electrographic, but not including epileptiform or other irritative discharges) in the 4 weeks prior to enrollment (individuals with premorbid idiopathic epilepsy are eligible to enroll under two conditions: a) if their pre-injury seizure frequency was less than once/month and they have had no more than 1 seizure/month since injury and b) if a clear provocation was present that would otherwise disqualify a subject, the subject can be enrolled, since these events would not be considered idiopathic),
* Prior exposure to AH post-TBI,
* Unwillingness to discontinue or change confounding psychotropic drugs prior to enrollment, OR
* Allergy or medical contraindication to AH and significant impairment of renal function (as evidenced by a calculated creatinine clearance of < 60 ml/min).

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2003-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T. Giacino, Ph.D., Principal Investigator — Spaulding Rehabilitation Hospital; John Whyte, MD, Ph.D., Principal Investigator — Moss Rehabilitation Research Institute
Locations (11):
- United States (8):
  - Braintree Rehabilitation Hospital, Braintree, Massachusetts
  - Methodist Rehabilitation Center, Jackson, Mississippi
  - Columbia University, New York, New York
  - Sunnyview Rehabilitation Hospital, Schenectady, New York
  - Charlotte Rehabilitation Center, Charlotte, North Carolina
  - Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - Bryn Mawr Rehabilitation Hospital, Malvern, Pennsylvania
  - Texas NeuroRehabilitation Center, Austin, Texas
- Hvidovre University Hospital, Hvidovre, Denmark
- Germany (2):
  - Neurologische Klinik Bad Aibling, Bad Aibling
  - Fachkrankenhaus Neresheim, Neresheim

REFERENCES:
- [Derived] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 23,2003 through March 15, 2010. Eleven rehabilitations centers in the USA (8) and Europe (3)
Groups:
- Placebo: Visually identical compound administered in the same manner (ie enterally) as the actual study drug.
Period: Overall Study
Arm/Group | Amantadine HCL | Placebo
Started | 87 | 97
Completed | 86 | 95
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amantadine HCL | Placebo | Total
Number analyzed (Participants) | 87 | 97 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 1 | 6
  Between 18 and 65 years | 82 | 96 | 178
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.5 (15.3) | 37.2 (15.4) | 36.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 64 | 69 | 133
Region of Enrollment [Number; unit: participants]
  United States | 61 | 73 | 134
  Denmark | 3 | 2 | 5
  Germany | 23 | 22 | 45

OUTCOME MEASURES:

1. Secondary Outcome: JFK Coma Recovery Scale-Revised: Neurobehavioral Status
Description: Measure of neurobehavioral function and clinical change for individuals with severe alterations of consciousness.
  Minimum score= 0; Maximum score= 23 (Higher scores are indicative of a higher-level of neurobehavioral function).
Time Frame: Week 4 (primary endpoint); Week 6 (post-washout)
Population: Analyses were conducted according to the ITT principle so that all 184 patients randomized were included for analysis. Imputation techniques were not undertaken since missing data were infrequent and unrelated to study outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Amantadine: Amantadine (200-400 mg/day)
- Placebo: Visually identical compound administered in the same manner (ie enterally) as the study drug.
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 87 | 97
units on a scale
  Week 4 (Primary endpoint) | 15.8 (6.1) | 14.2 (6.6)
  Week 6 (Post-washout) | 15.7 (6.3) | 15.1 (6.8)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; We will have 80% power to detect a one point difference in DRS score between the groups across the four week treatment window. With this sample size, we will be able to detect any unforeseen adverse events that have a prevalence of at least 2.5% in each group with 90% probability. With 92 patients per group we will be able to estimate the rate of adverse events to within ±10%; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis

2. Primary Outcome: Disability Rating Scale: Functional Status
Description: Measure of function after traumatic brain injury (TBI) intended to measure function from "coma to community." Minimum score= 0; Maximum score= 29 (High scores are indicative of greater degree of disability).
Time Frame: Randomization and weekly for 6 weeks. The primary study endpoint was week 4 and drug washout was week 6.
Population: Analyses were conducted according to the intention-to-treat principle. 184 subjects were randomized and included for analysis. Since missing data were infrequent and unrelated to the study outcome, imputation methods were not undertaken.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Amantadine | Placebo
Number analyzed (Participants) | 87 | 97
units on a scale
  Week 4 (Primary endpoint) | 17.3 (4.7) | 18.7 (4.5)
  Week 6 (Drug washout) | 17.1 (5.2) | 17.8 (5.3)
Statistical Analysis 1: Comparison: Amantadine vs Placebo; The planned sample size of 184 patients provided 80% power to detect a difference between the AH and placebo in the rate of Disability Rating Scale (DRS) score change of 0.3 points/week (1.22 DRS point mean difference by the end of the 4-week treatment interval). Two blinded interim analyses were conducted at 60 and 120 patients recruited using the O'Brien-Fleming boundary, with alpha levels of 0.0005 and 0.014. The final analysis used an alpha level of 0.045; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — The final analysis used a significance level of 0.045; Final analysis adjusted for early v. late enrollment relative to date of injury, baseline CRS-R rating category (MCS vs. VS), and site; Slope = -0.24, 95% CI [-0.41 to -0.07], Standard Error of Mean 0.088

ADVERSE EVENTS:
Arm/Group | Amantadine HCL | Placebo
Serious Adverse Events (participants affected / at risk) | 15/87 | 19/97
Other Adverse Events (participants affected / at risk) | 54/87 | 51/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine HCL (N=87) | Placebo (N=97)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 3 (3) | 2 (2)
Intracranial Hemorrage (Nervous system disorders) | 0 (0) | 1 (1)
Other Neurologic (Nervous system disorders) | 1 (1) | 1 (1) — Bilateral subdural fluid collection, arm and head tremor
Hypoarousal/Lethargy/Somnolence (Psychiatric disorders) | 0 (0) | 1 (1)
Autonomic Storm (Nervous system disorders) | 0 (0) | 1 (1)
Other Gastrointestinal Problems (Gastrointestinal disorders) | 2 (2) | 3 (3) — GI bleeding, gastritis, bowel obstruction, colon carcinoma, peritonitis
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 5 (5)
General Medical Problems (General disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Other Abnormal Laboratory (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Anemia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amantadine HCL (N=87) | Placebo (N=97)
Hypertonia / Spasticity (Musculoskeletal and connective tissue disorders) | 18 (21) | 14 (18)
Insomnia / Sleep Disturbance (General disorders) | 12 (14) | 14 (15)
Agitation / Aggression (Psychiatric disorders) | 12 (16) | 11 (14)
Infections (Infections and infestations) | 10 (14) | 15 (16) — Does not include urinary tract infection
Urinary tract infection (Renal and urinary disorders) | 13 (15) | 12 (13)
General Medical Problems (General disorders) | 9 (10) | 11 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less